CLINICAL TRIAL: NCT00148382
Title: Randomized, Double Blind, Parallel Group, Repeat Dose Pharmacokinetic and Pharmacodynamic Study of Four Doses of ATL-962 (40mg, 80mg, 120mg 240mg) in Otherwise-Healthy Obese Volunteers
Brief Title: Study of the Blood Levels and Effects of ATL-962 on Fat Excretion in Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alizyme (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATL-962/191/CL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Obesity
Keywords: Obesity; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Obesity | interventions — cetilistat

INTERVENTIONS:
Drug: ATL-962

SUMMARY:
The purpose of this study is to investigate the amount of metabolites of ATL-962 in the blood and to investigate the effect of ATL-962 on the amount of fat that is excreted in the faeces in subjects who are obese

DETAILED DESCRIPTION:
Obesity is a significant and increasing clinical problem. There is a need for effective therapeutic agents to help people reduce weight. ATL-962 is a lipase inhibitor which could reduce the amount of fat absorbed from a person's diet, leading to weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* Obese, otherwise-healthy subjects
* Body mass index 30-45kg/m2

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Any drug treatment within 2 weeks of commencement of dosing in this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2005-04; Study Completion 2005-07

PRIMARY OUTCOMES:
Pharmacokinetics of metabolites of ATL-962

SECONDARY OUTCOMES:
Effect of ATL-962 on faecal fat excretion
Safety and tolerability of ATL-962

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Galitz, Principal Investigator — SFBCI
Locations (1):
- SFBCI, Miami, Florida, United States